CLINICAL TRIAL: NCT04563702
Title: A Phase 1 Open-Label, Dose-Ranging Trial to Determine the Safety and Immunogenicity of an Adenoviral-Vector Based Vaccine (VXA-CoV2-1) Expressing a SARS-CoV-2 Antigen and dsRNA Adjuvant Administered Orally to Healthy Adult Volunteers VXA-CoV2-1.1-S Boost Substudy: Boost at 1 Year Post Initial Vaccination With an Adenoviral-Vector Based Vaccine VXA-CoV2-1.1-S Expressing a SARS-CoV-2 S Protein in a Subset of Subjects
Brief Title: Safety and Immunogenicity Trial of an Oral SARS-CoV-2 Vaccine (VXA-CoV2-1) for Prevention of COVID-19 in Healthy Adults and Boost (VXA-CoV2-1.1-S) at 1 Year Post Initial Vaccination in Subset of Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VXA-COV2-101
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2022-09

CONDITIONS: Covid19
Keywords: VXA-C0V2-1; Vaxart oral vaccine; tablet vaccine; VXA-C0V2-1.1; Boost
MeSH Terms: conditions — COVID-19 | interventions — VXA-CoV2-1 vaccine

STUDY DESIGN:
Intervention Model Description: Open-label, repeat dose, dose ranging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose VXA-CoV2-1 (Experimental): Low dose (1E10 I.U.) of VXA-CoV2-1 oral tableted vaccine dispensed at Day 1. A subset will also receive a second dose at Day 29
  Interventions: Biological: VXA-CoV2-1
- High Dose (Experimental): High Dose (1E11 I.U.) of VXA-CoV2-1 oral tableted vaccine dispensed at Day 1
  Interventions: Biological: VXA-CoV2-1

INTERVENTIONS:
Biological: VXA-CoV2-1 — non replicating Ad5 adjuvanted oral tableted vaccine

SUMMARY:
VXA-CoV2-1 is a non-replicating Ad5 vector adjuvanted oral tableted vaccine being developed to prevent COVID-19, the disease resulting from Severe Acute Respiratory Syndrome coronavirus (SARS-CoV-2) infection. The study is designed to evaluate the safety and immunogenicity of VXA-CoV2-1 vaccine with repeat dosing at multiple dose levels. Safety and immunogenicity will be evaluated for up to 12 months after the second dose of VXA-CoV2-1.

DETAILED DESCRIPTION:
This is an open-label, dose-ranging trial to determine the safety and immunogenicity of an orally administered adenoviral-vector based vaccine (VXA-COV2-1) expressing a SARS-CoV-2 antigen and dsRNA adjuvant. Post screening activities, healthy adult volunteers aged 18 - 54 yrs old, inclusive, will be enrolled into the study. Participants will receive an oral dose of vaccine at Days 1 and a subject will also receive a second dose at Day 29; total study period will last ~ 2 months during the active phase, with a total 12 month safety follow-up period post last vaccination. Safety, reactogenicity and immunogenicity assessments will be performed at set times during the study active and follow-up periods. Subjects will be monitored for symptoms of COVID-19 throughout the duration of the study follow-up period.

Approximately 10 healthy male and female adult volunteers 18 to 54 years old who were enrolled in the main study will be included in a boost extension substudy for an additional 12 months from dosing for a total participation period of 24-25 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 to 54 years, inclusive.
2. Negative for SARS-CoV-2 infection at the time of screening
3. In generally good health, without significant medical illness
4. Demonstrates comprehension of the protocol procedures and is able to provide written informed consent.
5. Available for all planned visits and willing to complete all protocol defined procedures and assessments
6. Body mass index between 17 and 30 kg/m2 at screening.
7. Female subjects must have a negative pregnancy test at screening and before each vaccination and fulfill an acceptable method of birth control (per protocol)

Exclusion Criteria:

1. Known previous exposure to SARS-CoV-2 or receipt of an investigational product for the prevention or treatment of COVID-19, middle east respiratory syndrome (MERS), or severe acute respiratory syndrome (SARS).
2. Is in a current occupation with high risk of exposure to SARS-CoV-2
3. Individuals with the following underlying medical conditions who are at higher risk (or might be at higher risk) of severe illness from COVID-19 per the CDC's guidance
4. Donation or use of blood or blood products within 4 weeks prior to vaccination or planned donation during the study period.
5. Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic.
6. Any condition that resulted in the absence or removal of the spleen.
7. Positive HIV, HBsAg or HCV tests at the screening visit.
8. Stool sample with occult blood at screening.
9. Use of antiviral medications, including anti-retrovirals, or any prescriptive medications for the prevention of COVID-19 within 7 days before vaccination
10. Use of antibiotics, proton pump inhibitors, H2 blockers or antacids or medications known to affect the immune function within 7 to 14 days before vaccination
11. Regular use of nonsteroidal anti-inflammatory drugs, sulfonylureas, and angiotensin II blockers within 7 days before vaccination
12. Acute disease within 72 hours prior to vaccination defined as the presence of a moderate or severe illness
13. History of drug, alcohol or chemical abuse within 1 year of screening or positive urine drug screen for drugs of abuse at screening
14. History of hypersensitivity or allergic reaction to any component of the investigational vaccine
15. Administration of any investigational vaccine, drug or device within 8 weeks preceding vaccination
16. Any other condition that in the clinical judgment of the investigator would jeopardize the safety or rights of a subject participating in the trial, would render the subject unable to comply with the protocol or would interfere with the evaluation of the study endpoints.

    For subjects being re-evaluated for participation in the VXA-CoV2-1.1-S boost substudy the following will also be exclusionary:
17. Laboratory values outside the range of normal for platelet counts and the following coagulation tests: PT/INR, aPTT, fibrinogen, and D-dimer.
18. Any of the following history or conditions that may lead to higher risk of clotting events and/or thrombocytopenia:

    e. Family or personal history of bleeding or thrombosis f. History of heparin-related thrombotic events, and/or receiving heparin treatments g. History of autoimmune or inflammatory disease h. Presence of any of the following conditions known to increase risk of thrombosis within 6 months prior to screening:
    * Recent surgery other than removal/biopsy of cutaneous lesions
    * Immobility (confined to bed or wheelchair for 3 or more successive days)
    * Head trauma with loss of consciousness or documented brain injury
    * Receipt of anticoagulants for prophylaxis of thrombosis
    * Recent clinically significant infection

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited symptoms of reactogenicity | Day 1 through Day 8 post each immunization
  Subject reported symptoms of local and systemic reactogenicity
Grade of solicited symptoms of reactogenicity | Day 1 through Day 8 post each immunization
  Subject reported symptoms of local and systemic reactogenicity
Frequency of unsolicited adverse events | Day 1 through Day 29 post each immunization
  Any adverse events observed or reported following vaccination
Grade of unsolicited adverse events | Day 1 through Day 29 post each immunization
  Any adverse events observed or reported following vaccination
Frequency of serious adverse events (SAEs) | Day 1 through Day 390
  Any adverse events reported following vaccination meeting definition of serious
Frequency of medically-attended adverse events (MAAEs) | Day 1 through Day 390
  Any adverse events reported following vaccination meeting definition of serious

SECONDARY OUTCOMES:
SARS-CoV-2 specific IgG/IgA | Day 1 through Day 390
  SARS-CoV-2 specific IgG/IgA by enzyme-linked immunosorbent assay (ELISA)
Neutralizing antibody titers to SARS-CoV-2 | Day 1 through Day 390
  serum based assay of Ab titers
Antigen-specific IgG/IgA antibody secreting (ASCs) | Day 1 through Day 44
  ASCs by ELISpot
Th1/Th2 polarization | Day 1 through Day 44
  Flow Cytometry

OTHER OUTCOMES:
SARS-CoV-2 specific IgG/IgA by enzyme-linked immunosorbent assay | Days 1, 29, 180 and 360
  MSD
Neutralizing antibody titers to SARS-CoV-2 | Days 1, 29, 180 and 360
  serum based assay of Ab titers
Antigen-specific IgG/IgA antibody secreting assays (ASCs) | Days 1 and Day 8
  ELISpot
Plasmablast immunophenotyping | Day 1 and Day 8
  Flow Cytometry
Detection of antigen S-specific IgA | Day 1 and Day 8
  Flow Cytometry
Detection of antigen S-specific IgA | Days 1, 29, 180, and 360
  Nasal swabs (SAM Device)
Detection of antigen S-specific IgA | Days 1, 29, 180, and 360
  Saliva
Cytof analysis of cell populations | Day 1 and Day 8
  Whole blood-based analysis
IFN-g production/IL-4 production by T cells | Day 1 and Day 8
  fresh whole blood/TrueCulture tube

CONTACTS AND LOCATIONS:
Overall Officials: James Cummings, MD, Study Director — Vaxart, Inc.
Locations (1):
- WCCT, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
A plan on how to share individual subject's outcomes will be defined within the next few months.

REFERENCES:
- [Derived] Langel SN, Johnson S, Martinez CI, Tedjakusuma SN, Peinovich N, Dora EG, Kuehl PJ, Irshad H, Barrett EG, Werts AD, Tucker SN. Adenovirus type 5 SARS-CoV-2 vaccines delivered orally or intranasally reduced disease severity and transmission in a hamster model. Sci Transl Med. 2022 Aug 17;14(658):eabn6868. doi: 10.1126/scitranslmed.abn6868. Epub 2022 Aug 17. PMID 35511920